CLINICAL TRIAL: NCT02075333
Title: The Effects of Ingesting or Rinsing Sucrose and Sucralose Solutions on Self-control, Cognitive Performance, and Blood Glucose Level
Brief Title: The Effect of Ingesting or Rinsing Sucrose and Sucralose on Self-control, Cognitive Performance, and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Sugar Nutrition, UK (Unknown)
Responsible Party: Principal Investigator, Prof Louise Dye, Chair of Nutrition and Behaviour, University of Leeds
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SN - 0114
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Self-control; Cognitive Performance; Blood Glucose Response
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose (50g) (Active Comparator): A 381g blackcurrant drink (cordial and water) providing 50g of sucrose
  Interventions: Dietary Supplement: Ingestion of solution; Dietary Supplement: Rinising of solution
- Sucralose (0.92 g sugars) (Placebo Comparator): A 381g blackcurrant drink (cordial and water) providing 0.92g of natural sugars
  Interventions: Dietary Supplement: Ingestion of solution; Dietary Supplement: Rinising of solution

INTERVENTIONS:
Dietary Supplement: Ingestion of solution — Participants will ingest the solution
Dietary Supplement: Rinising of solution — Participants rinse the solution in the oral cavity

SUMMARY:
The purpose of this study is to examine the effects of ingesting or mouth rinsing a sucrose (carbohydrate) versus a sucralose (carbohydrate-free) drink on self control, cognitive performance, and blood glucose level.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18 - 29 kg/m2

Exclusion Criteria:

* Dementia
* Depression
* Type 2 diabetes
* Phenylketonuria
* Intake of medication known to affect glucose metabolism
* Fasting blood glucose > 7.8 mmol/L

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose change from baseline following rinsing or ingesting sucrose or sucralose solutions | - 30, -15, - 5, + 5, + 10, + 20, + 30, + 40 minutes relative to rinsing or ingestion of sucrose or sucralose solutions (each separated by 7 days in crossover manner)
  Change from baseline in capillary blood glucose (assessed by lancet fingerprick and YSI blood glucose analyser)

SECONDARY OUTCOMES:
Visual verbal learning and memory performance following self-control depletion | + 35 minutes post ingestion or rinsing of sucrose or sucralose solutions (each separated by 7 days in crossover manner)
  Visual verbal learning performance will be assessed by the Visual Verbal Learning Test (Rey, 1964) following a self-control depletion task and ingestion or rinsing of a sucrose or sucralose solution
Attention switching performance following self-control depletion | + 20 minutes post ingestion or rinsing of sucrose or sucralose solutions (each separated by 7 days in crossover manner)
  Attention switching performance will be assessed by a switch task (Rogers and Monsell, 1995) following a self-control depletion task and ingestion or rinsing of a sucrose or sucralose solution
Continuous blood glucose change from baseline following rinsing or ingesting sucrose or sucralose solutions | 24 hours preceding and during ingestion or rinsing of sucrose or sucralose solutions (each separated by 7 days in a crossover manner)
  A subgroup of 10 participants recruited into the study will be fitted with a continuous glucose monitoring device (CGMS, iPRO) the day preceding each of the test days to measure continuous interstitial blood glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Neil B Boyle, Principal Investigator — University of Leeds; Louise Dye, Study Chair — University of Leeds
Locations (1):
- Human Appetite Research Unit (University of Leeds), Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided